CLINICAL TRIAL: NCT06854328
Title: A Prospective, Single Arm, Open Label Trial, to Confirm Safety and Effectiveness of Prism, as an Adjunct to Standard of Care, in Adolescents With Post-Traumatic Stress Disorder (PTSD)
Brief Title: The Prism Conformity Trial for Post-Traumatic Stress Disorder in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GrayMatters Health Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP008
Record Dates: First submitted 2025-02-24; First posted 2025-03-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-02

CONDITIONS: Post-Traumatic Stress Disorder in Adolescence
Keywords: Neurofeedback; PTSD in adolescent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single arm (Experimental): Eligible participants diagnosed with PTSD will be recruited from the community and from local clinical programs. All subjects will undergo Prism neurofeedback training.
  Participants will complete 15 neurofeedback training sessions delivered twice per week, on non-consecutive days, over 8 consecutive weeks.
  Interventions: Device: Prism

INTERVENTIONS:
Device: Prism — Prism is using an amygdala-fMRI-guided model for processing EEG signals. The model, termed EEG fMRI pattern (EFP), uses several electrodes EEG-signal to produce a real time amygdala-EFP biomarker signal. GrayMatters' product, Prism, is used to train patients in downregulating the amygdala-derived-EFP biomarker during therapy sessions.

SUMMARY:
Prism is a software as a medical device (SaMD) to be prescribed by clinicians as an adjunct to the standard of care treatment of patients with PTSD. The Prism software device runs on a laptop using an EEG signal input (g).Nautilos PRO (K171669).

The primary objective of the study is to extend the use of the FDA cleared Prism for PTSD (K222101) to an adolescent population and to confirm the safety of fifteen (15±3) EEG-NF training sessions using the Prism software in reducing PTSD-related symptoms in adolescents. The study aims to demonstrate the safety profile of Prism, having no device-related serious adverse events (SAEs), consistent with findings in the adult population, throughout the course of Prism treatment in an adolescent population.

DETAILED DESCRIPTION:
This study will be a Prospective, Single Arm, Open Label Trial, aiming to confirm the safety of the Prism system, adjunct to the standard of care, in adolescent subjects with PTSD.

Up to 45 subjects, but not less than 35, will be enrolled, and all will undergo Prism neurofeedback training. Participants will complete 15(±3) neurofeedback training sessions delivered twice per week, on non-consecutive days, over 8 consecutive weeks. A mid-training assessment will take place after 7 neurofeedback training sessions (week 4) and at the end of the training regimen (after completing the 15 ± 3 neurofeedback training - Week 8-9). A follow-up assessment will occur one (1) month after completing the last Prism training session.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 12 to 21 years.
2. Any gender.
3. Diagnosis of PTSD, established according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V).
4. ≥1 year since index trauma.
5. For candidate participants under 18 years old: Willingness and ability to provide assent, with the participant's legal guardian able and willing to provide informed consent for their study participation.
6. For candidate participants 18 years old and above: Willingness and ability to provide informed consent for their study participation.
7. English speaking, writing and reading.
8. Normal or corrected-to-normal vision and hearing.

Exclusion Criteria:

1. Have completed one or more full courses of trauma-focused therapy in the past (i.e., Eye Movement Desensitization and Reprocessing [EMDR], Prolong Exposure Therapy etc.), eligibility will be deemed upon the clinical judgement of the investigator.
2. Diagnosis for schizophrenia, schizoaffective disorder, schizophreniform disorder, Bipolar I disorder, or delusional disorder.
3. Any mood or anxiety disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5), that has been the primary focus of mental health treatment within the 6 months prior to screening, based on the clinical judgment of the site investigator.
4. Diagnosis of autism spectrum requiring substantial support, intellectual disability of mild severity at discretion of investigator.
5. Diagnosis of moderate or severe substance use disorder within the last 3 months of the screening visit (as defined in DSM-5-substance use disorder) or at the screening visit.
6. Current symptom level of moderate or severe ADHD (as defined in DSM-5 ADHD disorder) or at screening visit.
7. Any change in- or initiation of- psychotropic medications within the past 4 weeks. At the time of recruitment, subjects must have no intention of changing their medication or psychotherapy during the study duration.
8. Any suicidal behavior within the past 1 year (i.e., actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior), prior to screening and during the screening period.
9. Recent initiation (within the past 3 months) of cognitive-behavioral therapy or any evidence-based PTSD psychotherapy (Cognitive Processing Therapy [CPT], Prolonged Exposure [PE], Eye Movement Desensitization and Reprocessing [EMDR]). However, continuation of established maintenance supportive therapy will be permitted.
10. Any history of brain surgery, of penetrating, neurovascular, infectious, or other major brain injury, of epilepsy, or of other major neurological abnormality (including a history of traumatic brain injury [TBI] with loss of consciousness for more than 24 hours or posttraumatic amnesia for more than 7 days).
11. Any unstable medical condition, as per the clinical judgement of the investigator.
12. Enrollment in another interventional clinical study at screening or within 2 months prior to screening or intended enrollment within the duration of this study.
13. Female subjects who are pregnant, nursing, or who plan to become pregnant while in the trial.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Safety reporting | 1 month
  The primary objective of the study is to extend the use of the FDA cleared Prism for PTSD (K222101) to an adolescent population and to confirm the safety of Prism, by closely following and analyzing device-related serious adverse events. The success criterion is defined by no serious adverse event which is deemed as device-related during the study and one month after treatment ends.

SECONDARY OUTCOMES:
Proportion of participants improved in CAPS-5 | 9 weeks
  Assess the proportion of participants who demonstrate clinically meaningful improvement in the Clinician Administered PTSD Scale (CAPS-5) from Baseline to the post-training assessment visit (week 9)
Proportion of participants improved in PCL-5 | 9 weeks
  Assess the proportion of participants who demonstrate clinically meaningful improvement in the PTSD Checklist for DSM-5 (PCL-5) from Baseline to the post training assessment visit (week 9).

CONTACTS AND LOCATIONS:
Overall Officials: ADAR SHANI, Study Director — GrayMatters Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No